CLINICAL TRIAL: NCT06487052
Title: Evaluation of the Standard Catheter-directed Thrombolysis (SCDT) Effectiveness in Intermediate-High-Risk Pulmonary Embolism Patients
Brief Title: Evaluation of the Standard Catheter-directed Thrombolysis Effectiveness in Intermediate-High-Risk Pulmonary Embolism Patients
Acronym: ESCADlys-PE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Principal Investigator, Simakova Maria, Senior Researcher, Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1511-23
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Embolism Acute
Keywords: acute pulmonary embolism; catheter-directed thrombolysis; anticoagulant therapy
MeSH Terms: interventions — Fibrinolytic Agents

STUDY DESIGN:
Intervention Model Description: patients will be randomized into 2 parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Catheter-Directed Thrombolysis (Experimental): Local, standard catheter-directed thrombolysis with a total alteplase dose of 10 mg (for unilateral lesion) or 20 mg (for bilateral lesion) administered over 9 hours
  Interventions: Combination Product: Standard Catheter-Directed Low Dose Thrombolysis
- Standard Anticoagulation (Active Comparator): Therapy with UFH with targeted аPTT lasts for 24 hours (no more than 48 hours in total). Then the change to oral anticoagulants is performed.
  Interventions: Drug: Standard Anticoagulation

INTERVENTIONS:
Combination Product: Standard Catheter-Directed Low Dose Thrombolysis — Using femoral or jugular vein access the mechanical blood clots fragmentation by PigTail 6F catheter circular rotational movements. For unilateral thromboembolism, the PigTail catheter is positioned in the obstructed branch of the pulmonary artery, 1 mg of alteplase is injected as a bolus, followed by a micro-jet injection of 1 mg/hour. For bilateral thromboembolism, the PigTail catheter is positioned in the pulmonary trunk with a bolus of 2 mg alteplase followed by an infusion of 2 mg/hour. The total duration of infusion will be 9 hours, the total dose of alteplase will be 10 mg for unilateral lesions and 20 mg for bilateral lesions. During the alteplase infusion, unfractionated heparin is continued with a target activated partial thromboplastin time (aPTT) of 50 to 60 seconds. After completion of the procedure, UFH therapy is continued for 24 hours, followed by a change to oral anticoagulants.
  Arms: Standard Catheter-Directed Thrombolysis
Drug: Standard Anticoagulation — Therapy with UFH with targeted аPTT lasts for 24 hours (no more than 48 hours in total). Then the change to oral anticoagulants is performed
  Arms: Standard Anticoagulation

SUMMARY:
A single-center, open-label, randomized comparative study of two treatment strategies in patients with intermediate-high-risk acute pulmonary embolism (PE). Patients will be randomized in a 1:1 ratio to standard anticoagulant therapy or standard catheter-directed thrombolysis (SСDT) with a low dose of alteplase, followed by evaluation of short- and long-term efficacy and safety in each group

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Computed tomography angiography (CTA) - verified proximal (pulmonary trunk and/or main and/or lobar branches of the pulmonary artery) PE and symptom onset < 14 days prior
* Intermediate-high risk PE with a RV dysfunction (RV/LV diameter ratio >1 on TTE or CTA) and an elevated biomarker (hs-troponin or NT-proBNP) level
* Signed informed consent

Exclusion Criteria:

* High-risk pulmonary embolism
* Thrombus in the heart chambers on TTE
* Absolute contraindications for the use of thrombolytic therapy: history of hemorrhagic stroke or stroke of unknown etiology; ischemic stroke or transient ischemic attack within the last 6 months; extensive bleeding currently or within the previous 6 months, hemorrhagic diathesis; diseases of the central nervous system (including neoplasms, aneurysm, surgery on the brain or spinal cord); intracranial (including subarachnoid) hemorrhage currently or in history, suspicion of hemorrhagic stroke; severe uncontrolled arterial hypertension; major surgery or major trauma within the previous 3 months, recent traumatic brain injury; labor during the previous 10 days; severe liver diseases, including liver failure, cirrhosis, portal hypertension (including esophageal varices) and active hepatitis; bacterial endocarditis, pericarditis; acute pancreatitis; confirmed peptic ulcer of the stomach or duodenum within the last 3 months; arterial aneurysms, congenital anomalies of arteries/veins;
* Haemoglobin level < 70 g/L, platelet count ≤ 100 x 109
* Allergic to alteplase or UFH or contrast allergy
* Pregnant or breastfeeding
* Clinically significant malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
A decrease in the ratio of RV/LV diameters | 48 ± 6 hours
  A decrease in the ratio of RV/LV diameters by 20% or more from the initial value 48 ± 6 hours after initiation of therapy

SECONDARY OUTCOMES:
Mortality | 90 days
  Mortality
Cardiorespiratory decompensation or collapse | 7 days
  necessity of inotropic and vasopressor support; cardiac arrest or need for CPR; obstructive shock, placement on extracorporeal membrane oxygenation (ECMO), intubation, or initiation of non-invasive mechanical ventilation
Major bleeding events | 7 days
  International Society on Thrombosis and Hemostasis (ISTH) major bleeding
PE thrombus load reduction | 48 hours
  Qanadli score by CT-scan
The degree of residual pulmonary artery thrombosis with perfusion deficiency | 180 days
  The degree of residual pulmonary artery thrombosis with perfusion deficiency by CT-scan
Post-pulmonary embolism syndrome formation | 180 days
  The presence of symptomatic pulmonary artery residual thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- Almazov National Medical Research Centre, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Konstantinides SV, Meyer G, Becattini C, Bueno H, Geersing GJ, Harjola VP, Huisman MV, Humbert M, Jennings CS, Jimenez D, Kucher N, Lang IM, Lankeit M, Lorusso R, Mazzolai L, Meneveau N, Ni Ainle F, Prandoni P, Pruszczyk P, Righini M, Torbicki A, Van Belle E, Zamorano JL; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of acute pulmonary embolism developed in collaboration with the European Respiratory Society (ERS). Eur Heart J. 2020 Jan 21;41(4):543-603. doi: 10.1093/eurheartj/ehz405. No abstract available. PMID 31504429